CLINICAL TRIAL: NCT04977180
Title: Phase II Trial of Cardioprotective Prophylaxis With Combination of Beta Blocker and Angiotensin-Converting Enzyme Inhibitors During Intensive Chemotherapy for Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Cardioprotection in AML
Acronym: AML 001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Michael Keng, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSR210151
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: AML; Acute Myeloid Leukemia
Keywords: cardioprotection
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (beta blocker and ACE inhibitor) (Experimental): Participants will receive a beta blocker (either metoprolol or carvedilol) and an ACE inhibitor (lisinopril) at standard doses based on tolerance starting from when they start induction therapy for AML through 90 days after the first day of the last cycle of therapy that includes an anthracycline (whether that is in the induction, re-induction, or consolidation phase of treatment). If participants are unable to tolerate either beta blocker (e.g., heart rate is low at baseline or is lowered to an unsafe level with the beta blocker), no beta blocker may be administered as part of this study treatment. They will also undergo regular assessments via ECG/EKG and echocardiogram, and to measure troponin levels.
  Interventions: Drug: Cardioprotection
- Standard Clinical Care (No Intervention): Participants will receive standard clinical care, but will also undergo regular assessments via ECG/EKG and echocardiogram, and to measure troponin levels

INTERVENTIONS:
Drug: Cardioprotection — Preventive beta blocker (metoprolol or carvedilol) and an ACE inhibitor (lisinopril)
  Arms: Treatment arm (beta blocker and ACE inhibitor)

SUMMARY:
Patients with acute myeloid leukemia (AML) often receive a drug called daunorubicin. Daunorubicin is a type of drug called an anthracycline, which increases the risk of some damage to the heart. Beta blockers and angiotensin-converting enzyme inhibitors (ACEi) are two types of drugs that are often used (and are FDA approved) to treat the type of damage to the heart caused by anthracyclines. They have also been used in some populations to prevent this type of heart damage. In this study, participants will be randomly assigned to either preventively take a beta blocker and ACEi or not to receive these. The primary purpose of the study is to look at how often people in each group develop this type of heart damage. The study investigators will also collect data about your quality of life and other changes in your heart function.

Frequency and severity of anthracycline-induced cardiotoxicity among patients receiving acute myeloid leukemia (AML) chemotherapy is unknown. We hypothesize that up-titrating study agents to maximum tolerated dosage at the time of induction (starting treatment for AML) will prevent the development of systolic dysfunction as determined on serial echocardiography.

DETAILED DESCRIPTION:
Participants will know which group they are assigned to, and if someone in the group not receiving the preventive drugs needs these drugs for their clinical care, they will be able to receive them.

Participants in both groups will receive the standard clinical care medicines and lab tests for their AML. Everyone will have electrocardiograms (also called ECGs or EKGs) and echocardiograms before and at multiple timepoints during the study. They will also have a special blood test to see their levels of troponin, a protein that helps with muscle contractions in your heart. All participants will complete questionnaires at a few timepoints during the study to measure their quality of life. Participants in the preventive beta blocker and ACEi group will take these drugs when they're in the hospital and at home, keeping a diary of when they take it when they're at home.

The hypothesis of the study is that taking a beta blocker and ACEi during initial therapy for AML and through about 90 days after they last take an anthracycline will prevent the development of this heart problem.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to conducting any study-specific screening procedures.
2. Willing and able to understand the nature of this study and to comply with both the study as well as follow-up procedures for the duration of the study.
3. Age ≥ 18 years old with newly-diagnosed Acute Myeloid Leukemia (AML)
4. ECOG performance status must be ≤ 2
5. Planning to receive initial induction therapy containing an anthracycline for AML. Participants may have started initial induction therapy if anthracycline has not yet been administered.
6. Adequate organ function as evidenced by the following laboratory findings:

   1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) or < 3 x ULN for patients with Gilbert's Syndrome
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
   3. Creatinine clearance > 60 mL/min
7. Ability to take oral medication and a willingness to adhere to the beta blocker and lisinopril regimen
8. Echocardiogram demonstrating an ejection fraction ≥ 50% prior to the initiation of induction chemotherapy
9. For females of reproductive potential and males: Agree to abstain from sexual activity or use reliable contraception while undergoing treatment with chemotherapy and/or ACE inhibitors due to the risk of teratogenicity to the fetus.

Exclusion Criteria:

1. Ongoing use of any beta blocker, ACEi, or angiotensin II receptor agonist (ARB) at the time of pre-enrollment screening.
2. Uncontrolled, intercurrent illnesses including but not limited to symptomatic unstable angina pectoris, cardiac arrhythmias not well controlled with medications, myocardial infarction in the 6 months preceding registration or psychiatric illness/social situations that would limit compliance with study requirements as determined by the study personnel, all at the discretion of the treating oncologist.
3. Patient receiving concurrent investigational agents, or those who have received an investigational agent within one week of registration.

Exception - Participants may receive concurrent investigational agents, or have done so within one week of registration if:

* The side effects of the drug are well studied and well known AND
* The drug is not known to be cardioprotective or cardiotoxic

  4. Females who are pregnant or lactating.

  5. Life-threatening illnesses other than AML, uncontrolled medical conditions or organ system dysfunction that, in the investigator's opinion, could compromise the patient's safety or study outcomes.

  6. Active, untreated and/or severe infections as determined by the treating oncologist.

  7. History of hematopoietic stem cell transplant (HSCT) with active graft vs host disease, immunosuppression other than low-dose prednisone (≤ 5mg) or calcineurin inhibitors within the four weeks preceding registration

  8 Moderate or severe mitral or aortic valve disease, as determined by echocardiography

  9. Congestive heart failure as clinically diagnosed by treating oncologist at the time of presentation for induction chemotherapy, or documented diagnosed by a previous physician.

  10. History of (repaired or unrepaired) congenital heart disease that precludes recommendation for or administration of additional anthracyclines

  11. Significant liver disease, including cirrhosis or history of transplant or hepatorenal syndrome)

  12. Bradycardia (defined as baseline resting heart rate ≤ 60 beats per minute) or third degree atrioventricular heart block at presentation for induction chemotherapy.

  13. Baseline resting systolic blood pressure < 95mmHg at presentation for induction chemotherapy.

  14. Documented allergy to beta blockers or ACE inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | Baseline through 90 days after first day of last cycle of anthracycline (usually up to 6 months later)
  As determined by echocardiogram

SECONDARY OUTCOMES:
Congestive heart failure | Baseline through 90 days after first day of last cycle of anthracycline (usually up to 6 months later)
  As diagnosed by treating physician
Changes in quality of life | Baseline through 90 days after first day of last cycle of anthracycline (usually up to 6 months later)
  As measured by the FACT-Leu questionnaire
Global longitudinal strain | Baseline through 90 days after first day of last cycle of anthracycline (usually up to 6 months later)
  As measured by echocardiogram
Troponin levels | Baseline through 90 days after first day of last cycle of anthracycline (usually up to 6 months later)
  Frequency of elevation in troponin and average troponin

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keng, MD, Principal Investigator — UVA
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No